CLINICAL TRIAL: NCT00757783
Title: A Multicenter, Open-label, Randomized Study to Assess the Metabolics, Efficacy, and Safety of Once-daily Darunavir Versus Atazanavir in HIV-infected Treatment-naive Adult Patients
Brief Title: Changes in Triglyceride and Other Lipids (Levels of Fats Found in Blood) When Taking Darunavir Compared to Atazanavir in HIV-infected Patients That Have Never Received Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tibotec, Inc (Industry)
Collaborators: Tibotec Therapeutics, a Division of Ortho Biotech Products, L.P., USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR015439; TMC114HIV4023 (Other: Tibotec, Inc.)
Record Dates: First submitted 2008-09-19; First posted 2008-09-23 (Estimated); Results first posted 2010-09-10 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-11

CONDITIONS: HIV
Keywords: HIV; AIDS; Immunodeficiency Virus, Human; PREZISTA; darunavir; TMC114; Protease Inhibitor; Truvada; Atazanavir; REYATAZ; HIV Infections; Treatment Naïve
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections | interventions — Ritonavir; Darunavir; Emtricitabine; Atazanavir Sulfate

ARMS (2):
- darunavir (Experimental): darunavir 800 mg tablet once daily for 48 weeks,emtricitabine [FTC]/tenofovir [TDF] 200/300 mg tablet once daily for 48 weeks,ritonavir 100 mg capsule or tablet once daily for 48 weeks
  Interventions: Drug: ritonavir; Drug: darunavir; Drug: emtricitabine [FTC]/tenofovir [TDF]
- atazanavir (Experimental): atazanavir 300 mg capsule once daily for 48 weeks,emtricitabine [FTC]/tenofovir [TDF] 200/300 mg once daily for 48 weeks,ritonavir 100 mg capsule or tablet once daily for 48 weeks
  Interventions: Drug: ritonavir; Drug: emtricitabine [FTC]/tenofovir [TDF]; Drug: atazanavir

INTERVENTIONS:
Drug: ritonavir — 100 mg capsule or tablet once daily for 48 weeks
  Arms: darunavir
Drug: ritonavir — 100 mg capsule or tablet once daily for 48 weeks
  Arms: atazanavir
Drug: darunavir — 800 mg tablet once daily for 48 weeks
  Arms: darunavir
Drug: emtricitabine [FTC]/tenofovir [TDF] — 200/300 mg tablet once daily for 48 weeks
  Arms: darunavir
Drug: emtricitabine [FTC]/tenofovir [TDF] — 200/300 mg once daily for 48 weeks
  Arms: atazanavir
Drug: atazanavir — 300 mg capsule once daily for 48 weeks
  Arms: atazanavir

SUMMARY:
The purpose of this research study is to compare changes in triglyceride and other lipids (levels of fats found in the blood) from Baseline (Day 1) to Week 12 for darunavir/ritonavir 800/100 mg once daily versus atazanavir/ritonavir 300/100 mg once daily in combination with a fixed-dose background regimen consisting of emtricitabine [FTC]/tenofovir [TDF] 200/300 mg once daily). This study will also evaluate the safety (adverse events), effectiveness, and tolerability of darunavir/ritonavir and atazanivir/ritonavir over 48 weeks.

DETAILED DESCRIPTION:
The purpose of this study is to expand our understanding of the metabolic effects of darunavir/ritonavir (DRV/r) in HIV-infected patients. This is a phase 4, multicenter, open-label, randomized (study drug assigned by chance), comparative study designed to compare changes in lipid, glucose, and insulin parameters in HIV-infected, anti-retroviral (ARV) naive patients treated with DRV/r 800/100 mg once daily (QD) versus atazanavir/ritonavir (ATV/r) 300/100 mg QD in combination with a common background of emtricitabine (FTC)/ tenofovir (TDF) 200/300 mg QD. In addition, changes in inflammatory markers will be measured. A substudy of the parent study TMC114HIV4023 will evaluate insulin sensitivity and endothelial function in a subset of patients. The study will be conducted at approximately 16 study sites in the United States. Approximately 60 HIV-1 infected, treatment-naive adult patients will be enrolled in the study. Screening will take place during a 4-week period. At the baseline visit, eligible patients will be randomized in a 1:1 ratio to receive DRV/r 800/100 mg QD or ATV/r 300/100 mg QD administered in combination with a fixed-dose background regimen consisting of emtricitabine (FTC)/tenofovir (TDF) 200/300 mg once daily. The treatment period is 48 weeks. Study assessments will be performed at clinic visits at the end of weeks 4, 8, 12, 24, 36, and 48. The primary endpoint will be assessed at week 12. All patients will return for follow up visits 1 week and 4 weeks after the completion of study treatment. During the treatment period, the patient will be seen at regular visits during which the investigator will assess the patient's medical condition, any Adverse Events and study drug compliance. Laboratory evaluations for efficacy and safety will be done at regular visits as well as blood pressure monitoring. Up to twenty patients (evenly randomized to receive DRV/r or ATV/r) who meet additional entry criteria will be enrolled in the substudy. The study hypothesis is the change in triglycerides and other lipids from baseline to week 12 will be similar in the DRV/r arm versus the ATV/r arm. The substudy hypothesis is that DRV/r will not adversely affect insulin sensitivity or endothelial function during 12 weeks of therapy, and the change from baseline in insulin sensitivity and endothelial function will be similar in the DRV/r arm versus the ATV/r arm. During the treatment period, the patient will be seen at regular visits during which the investigator will assess the patient's medical condition, any Adverse Events and study drug compliance. Laboratory evaluations for efficacy and safety will be done at regular visits as well as blood pressure monitoring. Patients will be randomized in a 1:1 ratio to receive darunavir/ritonavir 800/100 mg once daily (QD) plus emtricitabine (FTC)/tenofovir (TDF) 200/300 mg QD or atazanavir/ritonavir 300/100 mg QD plus emtricitabine (FTC)/tenofovir (TDF) for 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 RNA of 1000 copies/mL or more
* No previous treatment with antiretroviral drugs for more than 10 days
* Demonstrated sensitivity [Fold Change (FC) = lower Clinical Cut Off (CCO)] to tenofovir, darunavir and atazanavir
* Demonstrated sensitivity to emtricitabine defined as absence of M184V/I mutation
* Any CD4 (Cluster of Differentiation 4) cell count

Exclusion Criteria:

* Body mass index >30 kg/m2
* Laboratory parameters as follows: fasting glucose >110 mg/dL, Low-Density Lipoprotein (LDL) cholesterol >130 mg/dL, triglycerides >200 mg/dL
* Presence of any currently active AIDS-defining illness
* Treatment for primary HIV infection or postexposure prophylaxis for HIV
* Patients with acute or chronic hepatitis A, B or C infection

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2008-10; Primary Completion 2009-08 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec, Inc. Clinical Trial, Study Director — Tibotec, Inc
Locations (15):
- United States (15):
  - Los Angeles, California
  - Glastonbury, Connecticut
  - Washington D.C., District of Columbia
  - Fort Lauderdale, Florida
  - Miami, Florida
  - Orlando, Florida
  - Indianapolis, Indiana
  - Boston, Massachusetts
  - Minneapolis, Minnesota
  - St Louis, Missouri
  - Hillsborough, New Jersey
  - New York, New York
  - Cincinnati, Ohio
  - Philadelphia, Pennsylvania
  - Dallas, Texas

REFERENCES:
- [Derived] Overton ET, Tebas P, Coate B, Ryan R, Perniciaro A, Dayaram YK, De La Rosa G, Baugh BP. Effects of once-daily darunavir/ritonavir versus atazanavir/ritonavir on insulin sensitivity in HIV-infected persons over 48 weeks: results of an exploratory substudy of METABOLIK, a phase 4, randomized trial. HIV Clin Trials. 2016 Mar;17(2):72-7. doi: 10.1080/15284336.2016.1141468. PMID 26917112
- [Derived] Gupta SK, Mi D, Liu Z, Saha C. Endothelial, inflammatory, coagulation, metabolic effects and safety of etravirine in HIV-uninfected volunteers. AIDS Patient Care STDS. 2011 Jun;25(6):327-31. doi: 10.1089/apc.2011.0011. Epub 2011 Apr 6. PMID 21470045

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 68 participants were enrolled in the study, and out of which 65 were treated.
Groups:
- Darunavir: Darunavir;emtricitabine [FTC]/tenofovir [TDF];ritonavir. 800 mg tablet once daily for 48 weeks;200/300 mg tablet once daily for 48 weeks;100 mg capsule or tablet once daily for 48 weeks.
- Atazanavir: atazanavir;emtricitabine [FTC]/tenofovir [TDF];ritonavir. 300 mg capsule once daily for 48 weeks;200/300 mg once daily for 48 weeks;100 mg capsule or tablet once daily for 48 weeks
Period: Overall Study
Arm/Group | Darunavir | Atazanavir
Started | 34 | 31
Completed | 29 | 25
Not Completed | 5 | 6
Not completed — Adverse Event | 0 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Other | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Darunavir | Atazanavir | Total
Number analyzed (Participants) | 34 | 31 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.9 (10.35) | 36.9 (11.66) | 36.4 (10.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 29 | 27 | 56
Region of Enrollment [Number; unit: participants]
  US | 34 | 31 | 65

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Fasting Triglyceride (TG) Levels in the Lipid Evaluable (LE) Set at Week12
Description: Observed values.
Time Frame: Baseline, Week 12
Population: The LE set consisted of all subjects in the PP analysis set who remained on study through Week 48 and had a fasting lipid assessment at baseline and at least once post first dose of DRV or ATV prior to or on the Week 48 visit. Here, 'n' signifies those participants evaluable for this measure at specified time points for each group, respectively.
Measure: Mean (Standard Deviation); unit: milligram per deciliters (mg/dL)
Arm/Group | Darunavir | Atazanavir
Number analyzed (Participants) | 28 | 27
milligram per deciliters (mg/dL)
  Baseline (n=28,27) | 113.7 (57.40) | 114.2 (84.05)
  Change at Week 12 (n=27,27) | 22.0 (62.72) | 8.1 (81.15)

2. Secondary Outcome: Change From Baseline in Total Cholesterol (TC) Levels in the LE Set at Week 12 and 48
Description: Observed Values
Time Frame: Baseline, Week 12 and 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Darunavir | Atazanavir
Number analyzed (Participants) | 28 | 27
mg/dL
  Baseline (n= 28, 27) | 141.8 (28.30) | 165.1 (29.93)
  Change at Week 12 (n= 27, 27) | 20.3 (30.48) | 4.6 (26.66)
  Change at Week 48 (n= 26, 22) | 22.3 (30.74) | 11.8 (31.93)

3. Secondary Outcome: Change From Baseline in Low Density Lipoprotein (LDL) Direct in the LE Set at Week 12 and 48.
Description: Observed Values
Time Frame: Baseline, Week 12 and 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Darunavir | Atazanavir
Number analyzed (Participants) | 28 | 27
mg/dL
  Baseline (n=28, 27) | 84.6 (21.93) | 100.2 (23.89)
  Change at Week 12 (n=27, 27) | 13.6 (25.12) | 9.6 (20.78)
  Change at Week 48 (n=26, 22) | 14.7 (25.91) | 13.9 (27.14)

4. Secondary Outcome: Change From Baseline in High Density Lipoprotein (HDL) in the LE Set at Week 12 and 48.
Description: Observed Values
Time Frame: Baseline, Week 12 and 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Darunavir | Atazanavir
Number analyzed (Participants) | 28 | 27
mg/dL
  Baseline (n=28,27) | 37.9 (13.36) | 45.0 (13.56)
  Change at Week 12 (n=27,27) | 6.6 (11.58) | 2.2 (8.74)
  Change at Week 48 (n=26,22) | 6.0 (7.43) | 3.7 (9.89)

5. Secondary Outcome: Change From Baseline in Apolipoprotein A1 in the LE Set at Week 12 and 48.
Description: Observed Values
Time Frame: Baseline, Week 12 and 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: grams per liters (g/L)
Arm/Group | Darunavir | Atazanavir
Number analyzed (Participants) | 28 | 27
grams per liters (g/L)
  Baseline (n=28,27) | 1.1 (0.26) | 1.3 (0.22)
  Change at Week 12 (n=27,27) | 0.1 (0.21) | -0.007 (0.18)
  Change at Week 48 (n=26,22) | 0.1 (0.16) | 0.0 (0.19)

6. Secondary Outcome: Change From Baseline in Apolipoprotein B in the LE Set at Week 12 and 48.
Description: Observed Values
Time Frame: Baseline, Week 12 and 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Darunavir | Atazanavir
Number analyzed (Participants) | 28 | 27
g/L
  Baseline (n=28,27) | 0.7 (0.19) | 0.8 (0.19)
  Change at Week 12 (n=27,27) | -0.004 (0.20) | -0.05 (0.16)
  Change at Week 48 (n=26,22) | 0.0 (0.21) | 0.0 (0.17)

7. Secondary Outcome: Change From Baseline in TC/HDL Ratio in the LE Set at Week 12 and 48.
Description: Participants TC and HDL was analyzed at Baseline and Week 12 and 48. Change from Baseline at Week 12 and 48 was calculated as ratio using observed values.
Time Frame: Baseline, Week 12 and 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Darunavir | Atazanavir
Number analyzed (Participants) | 28 | 27
ratio
  Baseline (n=28,27) | 4.1 (1.14) | 3.9 (1.02)
  Change at Week 12 (n=27,27) | -0.1 (0.91) | -0.1 (0.67)
  Change at Week 48 (n=26,22) | 0.1 (1.06) | -0.1 (0.75)

8. Secondary Outcome: Change From Baseline in Glucose at Week 12 and 48.
Description: Participants glucose level was analyzed at Baseline and Week 12 and 48. Change from Baseline at Week 12 and 48 was reported.
Time Frame: Baseline, Week 12 and 48
Population: Intent-to-treat (ITT) population included participants who remained on study through Week 48 and had an assessment at baseline and at least once post first dose of DRV or ATV prior to or on the Week 48 visit. 'N'=participants evaluable for this measure and 'n'=participants evaluable for this outcome measure at specified time points for each group.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Darunavir | Atazanavir
Number analyzed (Participants) | 33 | 30
mg/dL
  Baseline (n=33,30) | 88.5 (12.37) | 89.7 (10.84)
  Change at Week 12 (n=30,29) | 1.5 (12.52) | 5.8 (14.55)
  Change at Week 48 (n=28,24) | 2.8 (9.10) | 6.4 (22.07)

9. Secondary Outcome: Change From Baseline in Insulin at Week 12 and 48.
Description: Participants insulin was analyzed at Baseline and Week 12 and 48 and change from Baseline at Week 12 and 48 were reported.
Time Frame: Baseline, Week 12 and 48
Population: The ITT population included participants who remained on study through Week 48 and had an assessment at baseline and at least once post first dose of DRV or ATV prior to or on the Week 48 visit. 'N'=participants evaluable for this measure and 'n'=participants evaluable for this outcome measure at specified time points for each group, respectively.
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Darunavir | Atazanavir
Number analyzed (Participants) | 33 | 30
IU/mL
  Baseline (n=33,30) | 5.96 (5.566) | 8.59 (14.278)
  Change at Week 12 (n=30,29) | -1.07 (4.970) | 0.70 (18.790)
  Change at Week 48 (n=28,24) | 0.95 (6.006) | -2.88 (16.731)

10. Secondary Outcome: Change From Baseline in Homeostasis Model Assessment-Insulin Resistance (HOMA-IR) at Week 12 and 48.
Description: Participants homeostasis model assessment-insulin resistance (HOMA-IR) were observed and change from Baseline were reported. HOMA-IR score was calculated as: (fasting plasma glucose*fasting serum insulin)/22.5. Low HOMA IR values indicate high insulin sensitivity and high HOMA IR values indicate low insulin sensitivity (insulin resistance).
Time Frame: Baseline, Week 12 and 48
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: HOMA-IR score
Arm/Group | Darunavir | Atazanavir
Number analyzed (Participants) | 27 | 22
HOMA-IR score
  Baseline (n=27,22) | 1.624 (1.6962) | 2.943 (6.0204)
  Change at Week 12 (n=20,21) | -0.483 (2.0243) | 0.105 (7.5121)
  Change at Week 48 (n=19,14) | 0.035 (2.2580) | -1.236 (8.0114)

11. Secondary Outcome: Antiviral Activity, Human Immunodeficiency Virus Type 1 (HIV-1) RNA.
Description: Number of Participants with antiviral activity, human immunodeficiency virus Type 1 (HIV-1) RNA less than (<) 50 copies per milliliters (copies/mL) or < 400 copies/mL.
Time Frame: Week 12 and 48
Population: The ITT population included participants who remained on study through Week 48 and had an assessment at baseline and at least once post first dose of DRV or ATV prior to or on the Week 48 visit.
Measure: Number; unit: number of participants
Arm/Group | Darunavir | Atazanavir
Number analyzed (Participants) | 34 | 31
number of participants
  Week12: HIV-1 RNA Less Than (<) 50 copies/mL | 13 | 19
  Week 12: HIV-1 RNA < 400 copies/mL | 28 | 29
  Week 48: HIV-1 RNA < 50 copies/mL | 25 | 22
  Week 48: HIV-1 RNA < 400 copies/mL | 28 | 24

12. Secondary Outcome: Number of Participants With Antiviral Activity, HIV-1 RNA, Missing Values as Treatment Failure (M=F)
Description: Number of participants with antiviral activity, HIV-1 RNA, missing values as treatment failure (Missing = Failure) were observed.
Time Frame: Week 12 and 48
Population: as for outcome 11
Measure: Number; unit: number of participants
Arm/Group | Darunavir | Atazanavir
Number analyzed (Participants) | 34 | 31
number of participants
  Week 12: HIV-1 RNA Less Than (<) 50 copies/mL | 13 | 19
  Week 12: HIV-1 RNA < 400 copies/mL | 28 | 28
  Week 48: HIV-1 RNA < 50 copies/mL | 25 | 22
  Week 48: HIV-1 RNA < 400 copies/mL | 28 | 24

13. Secondary Outcome: Change From Baseline in HIV-1 RNA Viral Load at Week 12 and 48.
Description: the HIV-1 RNA viral load was calculated using Log Base 10 transformed HIV-1 RNA observed values.
Time Frame: Baseline, Week 12 and 48
Population: The ITT population included participants who remained on study through Week 48 and had an assessment at baseline and at least once post first dose of DRV or ATV prior to or on the Week 48 visit. Here, 'n' signifies those participants evaluable for this measure at specified time points for each group, respectively.
Measure: Mean (Standard Deviation); unit: Log10 HIV RNA
Arm/Group | Darunavir | Atazanavir
Number analyzed (Participants) | 34 | 31
Log10 HIV RNA
  Baseline (n=34,31) | 5.016 (0.7846) | 4.562 (0.6535)
  Change at Week 12 (n=32,30) | -2.955 (0.8081) | -2.605 (0.7035)
  Change at Week 48 (n=29,24) | -3.269 (0.8304) | -2.902 (0.6620)

14. Secondary Outcome: Change From Baseline in CD4 Cell Count at Week 12 and 48, Observed Values.
Description: Participants' Cluster of Differentiation (CD) 4 Cell Count were at baseline and the change values at Week 12 and 48 were observed.
Time Frame: Baseline, Week 12 and 48
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: cells/micro L
Arm/Group | Darunavir | Atazanavir
Number analyzed (Participants) | 34 | 31
cells/micro L
  Baseline (n=34,31) | 268.3 (144.17) | 326.7 (174.13)
  Change at Week 12 (n=32,29) | 111.1 (97.25) | 68.3 (134.60)
  Change at Week 48 (n=29,25) | 217.4 (116.76) | 205.3 (153.54)

15. Secondary Outcome: Change From Baseline in Cluster of Differentiation (CD) 4 Cell Count at Week 12 and 48, Last Observation Carried Forward (LOCF).
Description: Participants' Cluster of Differentiation (CD) 4 Cell Count were observed at baseline and the change values at Week 12 and 48 was calculated using LOCF.
Time Frame: Baseline, Week 12 and 48
Population: The ITT population included participants who remained on study through Week 48 and had an assessment at baseline and at least once post first dose of DRV or ATV prior to or on the Week 48 visit. LOCF was applied. Here, 'n' signifies those participants evaluable for this measure at specified time points for each group, respectively.
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Darunavir | Atazanavir
Number analyzed (Participants) | 34 | 31
cells/uL
  Baseline (n=34,31) | 268.3 (144.17) | 326.7 (174.13)
  Change at Week 12 (n=34,31) | 103.4 (101.01) | 74.6 (132.49)
  Change at Week 48 (n=34,31) | 194.9 (139.68) | 187.7 (146.28)

16. Secondary Outcome: Change From Baseline in Cluster of Differentiation (CD) 4 Percent at Week 12 and 48, Last Observation Carried Forward (LOCF).
Description: Participants' Cluster of Differentiation (CD) 4 percent were observed at baseline and the change values at Week 12 and 48 was calculated using LOCF.
Time Frame: Baseline, Week 12 and 48
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: percentage of CD4 cells
Arm/Group | Darunavir | Atazanavir
Number analyzed (Participants) | 34 | 31
percentage of CD4 cells
  Baseline (n=34,31) | 18.6 (9.89) | 21.4 (9.25)
  Change at Week 12 (n=32,30) | 5.9 (6.02) | 4.5 (5.25)
  Change at Week 48 (n=29,25) | 9.6 (7.24) | 8.5 (5.51)

ADVERSE EVENTS:
Time Frame: Week 48
Description: Safety population included all participants who received at least one dose of study drug.
Arm/Group | Darunavir | Atazanavir
Serious Adverse Events (participants affected / at risk) | 5/31 | 5/29
Other Adverse Events (participants affected / at risk) | 28/31 | 25/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Darunavir (N=31) | Atazanavir (N=29)
Mitral Valve Incompetence (Cardiac disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Chest Pain (General disorders) | 0 | 1
Immune Reconstitution Syndrome (Immune system disorders) | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Fracture of Penis (Injury, poisoning and procedural complications) | 0 | 1
Muscle Strain (Injury, poisoning and procedural complications) | 1 | 0
Pneumonitis Chemical (Injury, poisoning and procedural complications) | 0 | 1
Blood Glucose Increased (Investigations) | 1 | 0
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Darunavir (N=31) | Atazanavir (N=29)
Neutropenia (Blood and lymphatic system disorders) | 2 | 2
Ocular Icterus (Eye disorders) | 0 | 5
Abdominal Distension (Gastrointestinal disorders) | 3 | 2
Abdominal Pain (Gastrointestinal disorders) | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 10 | 5
Dyspepsia (Gastrointestinal disorders) | 1 | 2
Flatulence (Gastrointestinal disorders) | 2 | 2
Nausea (Gastrointestinal disorders) | 8 | 2
Fatigue (General disorders) | 4 | 3
Pain (General disorders) | 2 | 0
Pyrexia (General disorders) | 4 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 4
Jaundice (Hepatobiliary disorders) | 0 | 3
Immune Reconstitution Syndrome (Immune system disorders) | 3 | 0
Seasonal Allergy (Immune system disorders) | 0 | 2
Folliculitis (Infections and infestations) | 0 | 2
Furuncle (Infections and infestations) | 0 | 2
Influenza (Infections and infestations) | 2 | 0
Oral Herpes (Infections and infestations) | 1 | 2
Tinea Pedis (Infections and infestations) | 2 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 2
Urinary Tract Infection (Infections and infestations) | 1 | 2
Blood Bilirubin Increased (Investigations) | 0 | 10
Blood Cholesterol Increased (Investigations) | 1 | 2
Low Density Lipoprotein Increased (Investigations) | 4 | 3
Neutrophil Count Decreased (Investigations) | 0 | 2
Weight Decreased (Investigations) | 2 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 3
Dizziness (Nervous system disorders) | 1 | 2
Headache (Nervous system disorders) | 2 | 2
Depression (Psychiatric disorders) | 1 | 6
Insomnia (Psychiatric disorders) | 1 | 3
Pollakiuria (Renal and urinary disorders) | 0 | 2
Penile Discharge (Reproductive system and breast disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Acne (Skin and subcutaneous tissue disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 1

LIMITATIONS AND CAVEATS:
65 subjects were enrolled/treated in the main study. 3 subjects were enrolled, randomized, not treated and excluded from analyses (n=68). An additional 18 subjects were enrolled in a substudy extension and excluded from the main analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If TTCA does not publish within 12 months after study conclusion or after TTCA confirms there will be no multicenter publication, Institution may publish their results from their site individually, provided TTCA has 60 day review for confidentiality and additional 60 day delay for patent application.